CLINICAL TRIAL: NCT06721013
Title: A Phase 1/2, Dose-finding Study Investigating the Safety and Efficacy of Pirtobrutinib in Adults With Immune Thrombocytopenia
Brief Title: A Study of Pirtobrutinib in Participants With Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 27294; J2N-MC-JZNZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — pirtobrutinib

STUDY DESIGN:
Intervention Model Description: Phase 1-Open label Sequential, Phase 2-Double-blind Parallel
Who Masked: Participant, Investigator
Masking Description: Phase 1-Open label, Phase 2-Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pirtobrutinib Phase 1 (Experimental): Pirtobrutinib administered orally
  Interventions: Drug: Pirtobrutinib
- Pirtobrutinib Phase 2 (Experimental): Pirtobrutinib administered orally
  Interventions: Drug: Pirtobrutinib
- Placebo Phase 2 (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally
  Arms: Pirtobrutinib Phase 1; Pirtobrutinib Phase 2
Drug: Placebo — Administered orally
  Arms: Placebo Phase 2

SUMMARY:
The purpose of the phase 1 part of this study is to evaluate how well pirtobrutinib is tolerated and what side effects may occur. The phase 2 part of the study will further investigate efficacy and safety of multiple pirtobrutinib dosages versus placebo.

The study drug will be administered orally in participants with Primary Immune Thrombocytopenia (ITP). Blood tests will be performed to check how much pirtobrutinib gets into the bloodstream and how long it takes the body to eliminate it.

The study will last up to approximately 16 weeks for phase 1 dose-escalation and 28 weeks for phase 2 dose-optimization, excluding screening.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of primary ITP, defined as isolated thrombocytopenia not associated with another known disease process
* Have documented history of response, defined as 2 or more platelet counts greater than or equal to 50,000/microliter (μL), to at least 1 prior line of therapy. Splenectomy is considered a line of therapy
* Have relapsed or treatment-resistant primary ITP, with no available therapies known to provide clinical benefit
* Have a platelet count less than 30,000/μL on 2 occasions more than 5 days apart in the 15 days before randomization
* Have adequate liver, renal, and hematologic functions as defined by a table
* Are willing to follow contraception requirements

Exclusion Criteria:

* Have a history of any thrombotic or embolic event within 12 months before screening
* Had a transfusion with blood or blood products or plasmapheresis within 14 days (Phase 1) or within 28 days (Phase 2) of randomization
* Have significant cardiovascular disease
* Have a diagnosis or history of hematologic malignancy
* Have hepatitis B virus (HBV) defined as positive for antigen of hepatitis B (HBsAg) or polymerase chain reaction (PCR) positive for HBV deoxyribonucleic acid (DNA)
* Have hepatitis C virus (HCV) defined as positive for anti-HCV antibodies and PCR positive for HCV ribonucleic acid (RNA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1-Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline Up to Week 4
  A summary of TEAEs and SAEs regardless of causality, will be reported in the Reported Adverse Events module
Phase 1-Dose Limiting Toxicity (DLT) of Pirtobrutinib | Baseline Up to Week 4
  DLTs of Pirtobrutinib
Phase 1-Number of Participants with Treatment-Related Adverse Events as Assessed by Vital Signs: Blood Pressure, Pulse Rate, and Body Temperature | Baseline Up to Week 16
  Blood Pressure, Pulse Rate, and Body Temperature
Phase 1-Number of Participants with Treatment-Related Adverse Events as Assessed by Clinical Lab Tests: Hematology, Clinical Chemistry, Urinalysis, Pregnancy, Hepatitis Serology and Cytomegalovirus (CMV) | Baseline Up to Week 16
  Hematology, Clinical Chemistry, Urinalysis, Pregnancy, Hepatitis Serology and Cytomegalovirus (CMV)
Phase 1-Number of Participants with Treatment-Related Adverse Events as Assessed by Electrocardiograms (ECGs): ECG QT Interval | Baseline Up to Week 16
  ECG QT Interval
Phase 2-Efficacy of Pirtobrutinib Versus Placebo | Baseline Up to Week 24
  Stable platelet response rate is defined as the proportion of participants achieving platelet count of greater than or equal to 50 thousand per microliter (k/μL) and on at least 4 of the 6 consecutive biweekly visits between weeks 14 and 24 in the absence of rescue therapy and prohibited concomitant medication that may impact efficacy

SECONDARY OUTCOMES:
Phase 1-Preliminary Efficacy of Pirtobrutinib | Day 1 Up to Week 12
  Platelet response rate defined as proportion of participants who achieve at least 2 consecutive platelet counts of greater than or equal to 50 k/μL and an increase from baseline of greater than or equal to 20 k/μL to any time during treatment without the use of rescue medication within 4 weeks prior to the latest elevated platelet count.
Phase 1-Evaluate the Extent of Disease Control | Day 1 Up to Week 12
  Number of cumulative weeks with platelet counts greater than or equal to 50 k/μL by Week 12
Phase 1: Pharmacokinetics (PK) of Pirtobrutinib | Baseline Up to Week 16
  PK: Plasma Concentrations of Pirtobrutinib
Phase 2-Assess Additional Efficacy of Pirtobrutinib Versus Placebo | Week 14 Up to Week 24
  Platelet response rate is defined as the proportion of participants with greater than or equal to 2 consecutive platelet counts greater than or equal to 50 k/μL and an increase of platelet count of greater than or equal to 20 k/μL from baseline to any time during treatment or follow-up without the use of rescue medication or prohibited concomitant medication that may impact efficacy within 4 weeks prior to the latest elevated platelet count
Phase 2-Evaluate the Extent of Disease Control of Pirtobrutinib Versus Placebo | Baseline Up to Week 24
  Number of cumulative weeks with platelet counts greater than or equal to 50 k/μL and greater than or equal to 100 k/μL
Phase 2-Describe the Use of Rescue Medications of Pirtobrutinib Versus Placebo | Baseline Up to Week 24
  Proportion of participants requiring rescue therapy
Phase 2-Describe the PK of Pirtobrutinib | Week 16 Up to Week 40
  PK: Plasma Concentrations of Pirtobrutinib

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (45):
- United States (11):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford University, Stanford, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami Hospital and Clinics Sylvester Comprehensive Cancer Center, Miami, Florida
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Ochsner Medical Center - New Orleans, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Clinical Research Alliance, Westbury, New York
  - Texas Oncology-Central Austin, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology Gulf Coast, The Woodlands, Texas
- China (4):
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - Qilu Hospital of Shandong University, Jinan
  - Hematology Hospital of the Chinese Academy of Medical Sciences, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
- OUH, Odense C, Denmark
- France (3):
  - Hôpital Henri Mondor, Créteil
  - CHU Dijon - Hopital du Bocage, Dijon
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac
- Italy (4):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI), Trieste
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Sykehuset Ostfold, Kalnes, Grålum
  - St. Olavs Hospital Hf, Universitetssykehuset i Trondheim, Trondheim
- Poland (5):
  - Pratia Onkologia Katowice, Katowice
  - Pratia MCM Krakow, Krakow
  - Aidport sp z o.o., Skorzewo
  - MICS Centrum Medyczne Torun, Torun
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital General Universitario Morales Meseguer, Murcia
  - Clinica Universidad de Navarra, Pamplona
- United Kingdom (5):
  - Bristol Haematology and Oncology Centre, Bristol
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Royal London Hospital, London
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lilly Trials — https://trials.lilly.com/en-US/trial/558415